CLINICAL TRIAL: NCT00742976
Title: Effects of Insulin Detemir and NPH Insulin on Renal Handling of Sodium, Fluid Retention and Weight in Type 2 Diabetic Patients
Brief Title: Effects of Insulin Detemir and NPH Insulin on Renal Handling of Sodium, Fluid Retention, and Weight in Type 2 Diabetic Patients
Acronym: Le-Na
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Tonny Jensen, Dept. of Endocrinology; Rigshospitalet.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: EudraCT 2008-001602-16
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2008-06

CONDITIONS: Diabetes Type 2; Weight Gain
Keywords: Weight gain in insulin treated type 2 diabetes; extracellular volume; insulin treatment; sodium retention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Weight Gain; Hypernatremia | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 8 weeks of insulin Detemir, then cross over to 8 Weeks of Insulatard, then cross over to 1 week of Detemir
  Interventions: Drug: Insulin Detemir, Insulin Insulatard
- 2 (Active Comparator): 8 weeks of Insulin Insulatard, then cross over to 8 weeks of insulin Detemir, then crossover to 1 week of Insulin Insulatard
  Interventions: Drug: Insulin Detemir; Insulin Insulatard; Drug: Insulin Detemir, Insulin Insulatard

INTERVENTIONS:
Drug: Insulin Detemir; Insulin Insulatard — Dosage is individual but fixed in study period (if possible). Detemir is given once daily, Insulatard is given twice daily.
  Arms: 2
Drug: Insulin Detemir, Insulin Insulatard — Fixed doses in study period (if possible). Insulin Detemir once daily, Insulin Insulatard twice daily.

SUMMARY:
Hypothesis: Changing type 2 patients treatment from Insulin Insulatard to Insulin Detemir will increase their excretion of sodium in the urine and thereby decrease their extracellular volume and body weight. 24 patients are divided into 2 groups and their insulin treatment is shifted while their body composition, sodium excretion, weight and extracellular volume is monitored.

DETAILED DESCRIPTION:
Type 2 diabetic patients experience weight gain when receiving insulin treatment. There has been reports that the weight gain is less or absent when patients are treated with Insulin Detemir. Patients with diabetes have increased total body sodium and increased extracellular volume. We hypothesize that part of the weight gain seen is due to increase in extracellular volume and that the lesser weight gain seen in patients treated with Detemir is due to an lesser increase in extracellular volume. We believe that the cause of this difference is the different pharmacokinetic properties of insulin Detemir. Insulin Detemir i protein bound and is therefore not excreted in the kidneys. This may cause less sodium reabsorption, than with other insulins, and therefore less increase in extracellular volume.

We test this hypothesis by examining urinary sodium excretion, extracellular volume by GFR measurements, Body composition by DEXA scan, body weight, and 24 hour blood pressure.In patients that are changed from Insulin Insulatard to Insulin Detemir and back.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes according to WHO 1999 criteria for at least 3 month
* Insulin treated for at least 1 month
* BMI 25-40
* Age 18-80
* Hb1Ac < 10%

Exclusion Criteria:

* Hypertension not well regulated
* Serum creatinine > 130 micromol/l
* Non-diabetic kidney disease
* Disease that may cause invalid hgbA1c measurement
* Substance abuse
* Recent use of Detemir
* Pregnancy or risk of becoming pregnant
* Any condition that may disturb protocol adherence (language barrier etc) urinary albumin > 30 mg/24hours ( before screening)
* Use of drugs that may influence blood glucose (except oral antidiabetics)
* Use of drugs that may influence sodium balance,i.e diuretics ( tiazides accepted)
* Clinical significant disease that may influence outcome ( cancer etc)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
change in weight; change in extracellular volume | 17 weeks

SECONDARY OUTCOMES:
sodium excretion in urine, 24 hour blood pressure, body composition change,urine osmolality, urine albumin excretion, GFR, HbA1c, Blood lipid profile, NT-proBNP, plasma Albumin, Plasma metanephrines, aldosterone, active renin, angiotensin II | 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tonny Jensen, M.D MSci., Principal Investigator — Dept of Endocrinology at Rigshospitalet, Copenhagen.
Locations (1):
- Dept of Endocrinology, Rigshospitalet, Copenhagen, København Ø, Denmark

REFERENCES:
- [Derived] Hendriksen KV, Jensen T, Oturai P, Feldt-Rasmussen B. Effects of insulin detemir and NPH insulin on renal handling of sodium, fluid retention and weight in type 2 diabetic patients. Diabetologia. 2012 Jan;55(1):46-50. doi: 10.1007/s00125-011-2345-8. Epub 2011 Oct 16. PMID 22002075